CLINICAL TRIAL: NCT00134914
Title: Effects of Buprenorphine/Naloxone in Treating Opioid Dependent Individuals
Brief Title: Effects of Buprenorphine/Naloxone Administered in Different Ways For Treating Opioid Dependence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Eric C. Strain/Principal Investigator, Johns Hopkins University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NIDA-08045-4; R01-08045-4; DPMC
Record Dates: First submitted 2005-08-23; First posted 2005-08-25 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2008-07

CONDITIONS: Opioid-Related Disorders
Keywords: opiate dependence
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Buprenorphine — single doses given by sublingual and parenteral routes

SUMMARY:
Buprenorphine is a treatment for opioid dependence. Naloxone is given in addition to buprenorphine in order to limit the abuse potential that is commonly associated with buprenorphine. The purpose of this study is to examine the effects of buprenorphine/naloxone when given through different routes and at different doses.

DETAILED DESCRIPTION:
Buprenorphine, a mixed agonist-antagonist opioid (or partial agonist), is a safe and effective treatment for opioid dependence. However, there is concern that buprenorphine may be abused due to its high abuse potential. A sublingual buprenorphine/naloxone combination tablet may reduce the risk of abuse associated with buprenorphine alone. The purpose of this study is to characterize the effects of buprenorphine/naloxone in opioid-dependent individuals.

This study will last 10 weeks. Participants will stay in a residential research unit, and will be maintained on oral hydromorphone (10 mg). During twice-weekly experimental sessions, participants will be randomly assigned to receive either sublingual tablets, intramuscular injections, or a placebo. The 15 conditions studied will include: sublingual or intramuscular buprenorphine/naloxone (1/0.25 mg, 2/0.5 mg, 4/1 mg, 8/2 mg, and 16/4 mg), 0.25 mg of intramuscular naloxone (antagonist control), 10 mg of intramuscular hydromorphone (agonist control), sublingual and intramuscular buprenorphine (8 mg), and placebo.

ELIGIBILITY:
Inclusion Criteria:

* Currently opioid dependent
* In good health, as determined by a pre-participation medical examination
* Seeking and eligible for methadone maintenance or detoxification treatment

Exclusion Criteria:

* Significant medical or psychiatric illness, other than drug dependence

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 1996-08; Primary Completion 1998-04 (Actual); Study Completion 1998-05 (Actual)

PRIMARY OUTCOMES:
Opioid agonist rating | up to one day
opiate withdrawal | up to one day
physiologic measures | up to one day

CONTACTS AND LOCATIONS:
Overall Officials: Eric C. Strain, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University (BPRU) Bayview Campus, Baltimore, Maryland, United States

REFERENCES:
- [Result] Stoller KB, Bigelow GE, Walsh SL, Strain EC. Effects of buprenorphine/naloxone in opioid-dependent humans. Psychopharmacology (Berl). 2001 Mar;154(3):230-42. doi: 10.1007/s002130000637. PMID 11351930